CLINICAL TRIAL: NCT05806034
Title: Evaluation of Anterior Cruciate Ligament Tears Using Diffusion Tractography
Acronym: TRACTOLCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0098
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: ACL Injury; MRI; Tractography
Keywords: ACL Injury; MRI; tractography
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tractography MRI sequence protocol — tractography MRI sequence protocol does not require injection of contrast agent.

SUMMARY:
Knees injuries commonly affect the ACL. French current methodology is based on MRI focused on the knee with morphological sequences (T1, DP fat sat) allowing the study of ACL as follows: No lesion / Partial tear / Complete tear.

The treatment (kinesitherapy, surgery, no intervention) is defined taking into account several factors such as age, knee laxity, physical activity and outcome of the radiology analysis (partial or complete tear). However, if the classification is straightforward in case of complete tear, it is not possible to establish a quantitative impact on the ACL in case of partial tear. As a consequence, the investigators will analyze the anisotropy coefficient with diffusion tractography. Any patient who undergo a posttraumatic knee MRI at the CHU Amiens Picardie will have an appointment at the 3T "Signa" MRI that has the knee-centric diffusion tractography sequence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Patient referred for non-enhanced knee MRI for traumatism.
* Affiliation to a social security program,

Exclusion Criteria:

* Person under guardianship or curators,
* Any contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Anisotropy score after tractography MRI sequence | one day
  Anisotropy coefficient value is between 0 (isotropic medium) to 1 (fibrillar medium) .
  Anisotropy coefficient =0 is for total ACL rupture Anisotropy coefficient between 0 end 0.8 is for partial ACL rupture
Correlation between anisotropy coefficient and ACL lesion state | one year
  Anisotropy coefficient value is between 0 (isotropic medium) to 1 (fibrillar medium) .
  Anisotropy coefficient =0 is for total ACL rupture ACL lesion state are No lesion, Partial tear or Complete tear

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No